CLINICAL TRIAL: NCT03426020
Title: The Effect of Three Different Interventions on the Recovery Agitation and Delirium in the Pacu Pediatric Patients
Brief Title: The Effect of Premedication Type(Pharmalogical and Non Pharmalogical) on Delirium
Acronym: EDIRA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Reyhan Polat, Associate Profesor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 27/11/2017 43/20; Ministry of Health (Other: Diskapi Yildirim Beyazit Education and Research Hospital)
Record Dates: First submitted 2017-12-12; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2017-12

CONDITIONS: Emergence Agitation
Keywords: Premedication; Pediatric patients; Emergence agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Effect of pharmacologic or nonpharmacologic premedication on emergency agitation
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral midazolam (Demizolam®) (Active Comparator): To prevent emergence agitation patient premedicated by 0.5 mg oral midazolam At the end of sugery patients postoperatif emergence agitation evaluated by PAED(pediatric anesthesia emergence delirium scale).
  Interventions: Other: Oral midazolam
- Film http://www.animaturk.com/animasyon/suko-ameliyat-oluyor (Active Comparator): To prevent emergence agitation patient premedicated by watching a short movie (at URL: http://www.animaturk.com/animasyon/suko-ameliyat-oluyor ) At the end of sugery patients postoperatif emergence agitation evaluated by PAED(pediatric anesthesia emergence delirium scale).
  Interventions: Other: Film http://www.animaturk.com/animasyon/suko-ameliyat-oluyor
- Play game (PC fishing game) (Active Comparator): To prevent emergence agitation patient premedicated by playing a simple PC game (fishing game) At the end of sugery patients postoperatif emergence agitation evaluated PAED(pediatric anesthesia emergence delirium scale).
  Interventions: Other: Play game (PC fishing game)

INTERVENTIONS:
Other: Oral midazolam — 0.5 mg/kg oral midazolam administered 20 minutes before induction
  Other Names: Demizolam
  Arms: Oral midazolam (Demizolam®)
Other: Film http://www.animaturk.com/animasyon/suko-ameliyat-oluyor — patients will be watched a short movie (at URL: http://www.animaturk.com/animasyon/suko-ameliyat-oluyor ) 20 minutes before induction.
  Arms: Film http://www.animaturk.com/animasyon/suko-ameliyat-oluyor
Other: Play game (PC fishing game) — Patients will be played a simple PC game (a fishing game) 20 minutes before induction
  Arms: Play game (PC fishing game)

SUMMARY:
Compare the effects of pharmacologic and nonpharmacologic premedications on postoperative emergence delirium and preoperative anxiety, vital parameters, blood pressure, heart rate, SpO2, and pain at PACU 15 minutes after adenotonsillectomy .

DETAILED DESCRIPTION:
Compare the effects of

0.5 mg/kg oral midazolam,

watching film "Suko is being operated 'animation film (http://www.animaturk.com/animasyon/suko-ameliyat-oluyor.html#.Wd-YhFu0PIU) and

playing a game named "fishing games" on postoperative emergency delirium by PAED (post anestesic emergency delirium) scale at PACU at arrive and every 5 minutes for 15 minutes after adenotonsillectomy.

Investigators also evaluated "Basic and 20 minutes after pharmacologic and nonpharmacolgic premedications on participitans anxiety by Modified Yale Preoperative Anxiety Scale m-YPAS scores"

Pain evaluated by FLACC (behoviaral pain assesment scale),at arrive and every 5 minutes for 15 minutes after adenotonsillectomy.

Blood pressure(mmHg), heart rate(beat/min) and SpO2(%) measured and recorded at arrive and every 5 minutes for 15 minutes after adenotonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Pediatric patients
* Elective surgery
* Adenotonsillectomi

Exclusion Criteria:

* Cronicdesease
* Mental retarde
* Hearing and visual impaired
* Prematurite

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2018-02-20 (Estimated); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-06-10 (Estimated)

PRIMARY OUTCOMES:
Emergence agitation | Postoperative every 5 minutes for 15 minutes
  Emergence agitation will be evaluated by PAED (pediatric anesthesia emergence dellirium).The PAED scale consists of five behaviors, each of which is rated on a five-level scale with a score of zero to four. The scores are added to achieve a total scale score (maximum value is 20). The score above 12 is significant for post operative emergence agitation.

SECONDARY OUTCOMES:
preoperative anxiety | 20 minutea after premedications.
  Preoperative anxiety will be evaluated by Modified Yale Preoperative Anxiety Scale ( m-YPAS )scores. Range between 23 to 100. m-YPAS score above 30 is significant to patients anxiety.
Post operative pain | Postoperative every 5 minutes for 15 minutes
  Postoperative pain will be evaluated by behavioral pain scale FLACC(behavioral pain assesment scale). Each of the five categories (F) Face; (L) Legs; (A) Activity; (C) Cry; (C) Consolability is scored from 0-2, which results in a total score between zero and ten. 0 = Relaxed and comfortable.
  1 - 3 = mild discomfort 4 - 6 = moderate pain 7 - 10 = Severe discomfort or pain or both
Mean arteriel pressure | Postoperative every 5 minutes for15 minutes
  Mean arteriel pressure, will be measured. Mean blood pressurre range between 66 to 73 mm Hg is considered normal value. 20% increase in baseline value is considered significant.
Heart rate | Postoperative every 5 minutes for15 minutes.
  Heart rate range between 80 to 120 beats/minute is considered normal value. %20 percent increase in baseline value is considered significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Reyhan Polat, Ankara, Turkey (Türkiye)